CLINICAL TRIAL: NCT02455414
Title: Tracking Neurodegeneration in Early Wolfram Syndrome
Acronym: TRACK
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201301004; R01HD070855-02 (NIH)
Record Dates: First submitted 2015-03-05; First posted 2015-05-27 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Type 1 Diabetes; Diabetes Insipidus; Diabetes Mellitus; Wolfram Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Insipidus; Diabetes Mellitus; Wolfram Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A skin biopsy will be obtained from which the investigator will sequence all the exons and exon-intron junctions of the WFS1 gene. In some cases, the investigator will also sequence other genes related to Wolfram syndrome including WFS2, MANF, and Caspase-12. If the investigator doesn't find mutations in these genes, a whole-exome sequencing may be performed. The genetic test provided has the potential to create a uniquely-identifiable fingerprint that could possibly identify a participant.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Wolfram Syndrome Group: * Participant has confirmation of a WFS1 mutation OR
  * Both of the following conditions: diabetes mellitus requiring insulin and optic nerve atrophy diagnosed by a physician. Both conditions diabetes mellitus and optic nerve atrophy had to be diagnosed at age younger than 18 years old
- WFS Pre-symptomatic Sibling Group: * Has had genotyping
  * Willingness to share result of genotyping
  * Participant has confirmation of WFS1 (+/+) mutation but is asymptomatic.
- WFS Control Sibling Group: * Has had genotyping
  * Willingness to share result of genotyping
  * Patient has confirmation of NO WFS1 mutation (-/-) or confirmation as a carrier (+/- or -/+).
- T1DM Group: * Age within the 0-28 yrs age range of WS participant
  * Dx of T1 diabetes mellitus
- Healthy Control (HC) Group: • Age within the 0-28 yrs age range of WFS participants
- Proxy Group: Adult Biological parent(s), biological caregiver or non-biological caregiver of adult and minor participants in the any of the groups.

SUMMARY:
The goal of this study is to determine the pattern of early neurodegenerative changes in WFS (Wolfram Syndrome). The investigator will perform cross-sectional and longitudinal assessments of youth with WFS, targeting sensitive neural systems with quantified neuroimaging and behavioral measures. In addition, the investigator will establish the utility of a WFS severity rating scale (WFS Unified Rating Scale or WURS). Preliminary data support the feasibility of this approach and its potential to generate important new information about neurodevelopmental and neurodegenerative patterns in WFS. This work is necessary to position the field for future clinical trials to test interventions for WFS neurodegeneration. Ultimately, a better understanding of the trajectory of neurodegeneration in WFS and the development of effective interventions may be relevant to other more common neurodegenerative and endocrine (Type 1 and Type 2 diabetes) diseases in which ER stress has been implicated.

DETAILED DESCRIPTION:
Specific Aims: Wolfram syndrome (WFS) is a rare (1 in ~770,000) autosomal recessive genetic disease characterized by early childhood onset insulin dependent diabetes, optic nerve atrophy, vision and hearing loss, diabetes insipidus and neurodegeneration, resulting in death in middle adulthood, typically due to brainstem atrophy-induced respiratory failure 3. There are no interventions to slow or stop this devastating deterioration. However, much is known about the mechanisms underlying these effects. The causative gene (WFS1) was identified by the investigators group in 19984, and a number of loss-of-function mutations have been described 4-6. Cell 7 and animal models 8 have determined that WFS1 encodes an endoplasmic reticulum (ER) membrane-embedded protein called wolframin 9, and that mutant forms of the WSF1 protein lead to disturbances of ER calcium homeostasis, driving ER stress-mediated apoptosis 10-12. This process kills insulin producing pancreatic β-cells, leading to diabetes. WFS1 is also expressed throughout the brain, and cell death via ER stress is thought to underlie neurodegeneration in WFS 6,13, as well as being implicated in more common neurodegenerative and endocrine (Type 1 and Type 2 diabetes) diseases 14. Work in animal models of WFS is progressing rapidly towards the identification of viable interventions for the ER stress related cell death12. Some neurological features of the disease may be feasible to target and monitor in clinical trials, due to the fact that diabetes is already present when a patient is diagnosed with WFS. Unfortunately, there is limited information on the pattern of brain changes associated with WFS. Although clinical retrospective data suggest that neurological features occur late (15-30 yrs of age; Fig 10) in the disease process15,16, direct measurements (Preliminary Data) suggest that certain neurological abnormalities are present at the earliest time point assessed, suggesting altered neurodevelopment, whereas others follow a more neurodegenerative pattern. These distinctions are fundamentally new insights into this disease and may shape treatment, biomarker selection and the investigators understanding of the impact of ER stress on the developing brain. A better understanding of the neurodegenerative and neurodevelopmental changes in early WFS is a necessary first step towards being ready for future clinical trials. Thus, the primary goal of this proposal is to determine the pattern of brain alterations in WFS over time. Only by understanding the natural history of brain functional and structural changes in WFS will the investigator be prepared to evaluate any benefits of novel treatments. The investigator will perform cross-sectional and longitudinal assessments of youth with WFS, targeting sensitive neural systems with quantified neuroimaging and relevant behavioral measures. In addition, the investigator will validate a new WFS severity rating scale (WFS Unified Rating Scale or WURS), which will have utility in future multi-site or treatment studies. Preliminary data support the feasibility of this approach and its potential to generate important new information about neurologic patterns in WFS. A better understanding of the trajectory of ER stress-mediated brain changes in WFS may be relevant to other more common diseases. Specific aims follow:

1. To determine the pattern of neurologic impairment in WFS and its association with disease severity in a cross-sectional sample. The investigator hypothesizes that specific brain measures will be altered earlier and will associate more closely with overall disease severity than others in WFS. The investigator proposes that regional white matter microstructural integrity in the cerebellum, optic nerve area, brain stem volume, balance and possibly anxiety will distinguish individuals with early WFS from controls and will correlate with severity on a standardized rating scale. To test this hypothesis, the investigator will perform quantified neuroimaging, cognitive, motor, psychiatric, visual and auditory evaluations on individuals with WFS, preferentially recruiting those earlier in the disease process, (n=30; age 5 and older, within 10 years of diabetes onset) and on matched healthy controls (n=30) and controls with Type 1 Diabetes Mellitus (T1DM; n=30).
2. To determine the longitudinal pattern of neurologic deterioration in WFS. The investigator hypothesize that measures specified in Aim 1 will show detectable change, and that the most sensitive measures will show change in the early Wolfram patients compared to control groups. To test this hypothesis, WFS, T1DM and control participants will be re-assessed annually for 3 years. Variables of interest identified in cross-sectional analyses will be targeted and compared between groups and correlated with change in disease severity as measured with the investigators standardized rating scale.
3. To explore brain structure-function relationships within WFS. To determine if neuroimaging measures identified in Aims 1 and 2 have functional correlates, the investigator will explore how differences (cross-sectional data) or change (longitudinal data) in neuroimaging variables correlate with differences or change in selected functional measures. Such data would help build hypotheses about the neural underpinnings of functional changes in WFS. For example, the investigator speculates that the integrity of the brainstem and cerebellum will be related to gait and balance and that optic nerve area will be related to visual acuity.

ELIGIBILITY:
Wolfram Syndrome Group (WFS):

Inclusion Criteria:

* Participant has confirmation of a WFS1 mutation OR
* Both of the following conditions: diabetes mellitus requiring insulin and optic nerve atrophy diagnosed by a physician. Both conditions diabetes mellitus and optic nerve atrophy had to be diagnosed at age younger than 18 years old

Exclusion Criteria:

* Participant is unaware of their diagnosis.
* Inability of patient or guardian to understand informed consent.
* Advanced disease that makes traveling too problematic and/or uncomfortable for the patient and/or guardian, such as use of ventilator or inability to walk.

T1DM Group:

Inclusion criteria:

* Age within the 0-28 yrs age range of WS participant
* Dx of T1 diabetes mellitus

Exclusion criteria:

* Participant is unaware of their diagnosis.
* Inability of patient or guardian to understand informed consent.
* Diagnosis of any major neurological or medical condition.
* Chronic disease other than T1DM, well-controlled asthma, or Hashimoto's thyroiditis.
* Other current serious medical illness
* Co-morbid psychiatric illness: such as mania, mental retardation, or psychoactive drug dependence.
* Co-morbid neurological illness: stroke, seizure, major loss of consciousness, other brain trauma/surgery, or head injuries (i.e. near drowning), encephalitis, or hydrocephalus, blindness, deafness.
* Pre-maturity at birth >4 wks early (<36 wk term) w/ sequelae (e.g. on respirator at NICU)
* Contraindication to MRI scan (e.g. claustrophobia, metal implants, foreign bodies)
* Orthodontic braces. Full and top braces will exclude.

Healthy Control (HC) Group:

Inclusion criteria:

• Age within the 0-28 yrs age range of WFFS participants

Exclusion criteria:

* Inability of patient or guardian to understand informed consent.
* Dx of T1 diabetes mellitus
* Diagnosis of any major neurological or medical condition.
* Chronic disease other than well-controlled asthma, or Hashimoto's thyroiditis.
* Other current serious medical illness
* Co-morbid psychiatric illness: such as mania, mental retardation, or psychoactive drug dependence.
* Co-morbid neurological illness: stroke, seizure, major loss of consciousness, other brain trauma/surgery, or head injuries (i.e. near drowning), encephalitis, or hydrocephalus, blindness, deafness
* Pre-maturity at birth >4 wks early (<36 wk term) w/ sequelae (e.g. on respirator at NICU)
* Contraindication to MRI scan (e.g. claustrophobia, metal implants, foreign bodies)
* Orthodontic braces. Full and top braces will exclude. Bottom braces are ok (but the scan might not work out). Retainers are ok.

Proxy Group: Adult Biological parent(s), biological caregiver or non-biological caregiver of adult and minor participants in the any of the four groups.

Inclusion criteria:

• Biological or non-biological parent/caregiver (proxy) of a participant.

Exclusion criteria:

• Proxy is unaware of the participant's diagnosis (as it applies).

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Age, gender and handedness matched participants between the age of 1 day to no upper limit.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-04; Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Change in regional brain volume | annually for 5 years
  MRI measures of regional brain volumes over time

SECONDARY OUTCOMES:
Change in disease severity score | annually for 5 years
  WURS physical severity score over time

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Hershey, PhD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Bischoff AN, Reiersen AM, Buttlaire A, Al-Lozi A, Doty T, Marshall BA, Hershey T; Washington University Wolfram Syndrome Research Group. Selective cognitive and psychiatric manifestations in Wolfram Syndrome. Orphanet J Rare Dis. 2015 May 30;10:66. doi: 10.1186/s13023-015-0282-1. PMID 26025012